CLINICAL TRIAL: NCT06985992
Title: The Efficacy of Intrathecal Morphine Versus Intrathecal Morphine-Dexamethasone Combination in Cesarean Delivery: A Prospective Randomized Double-Blind Clinical Trial
Brief Title: The Efficacy of Intrathecal Morphine Versus Intrathecal Morphine-Dexamethasone Combination in Cesarean Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Nurettin KURT, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/04-05
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Caesarean Section
Keywords: Caesarean section; morphine; dexamethasone; nausea-vomiting; postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Spinal anesthesia will be administered to 120 pregnant patients scheduled for elective cesarean section, using either a combination of 2 mL (10 mg) bupivacaine, 0.1 mL (100 mcg) morphine, and 0.5 mL saline, or a combination of 2 mL (10 mg) bupivacaine, 0.1 mL (100 mcg) morphine, and 0.5 mL (2 mg) dexamethasone, depending on the group to which they are randomized.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group morfin (Active Comparator): Group Morphine: Spinal anesthesia will be applied to patients who will undergo caesarean section using a combination of 2 ml (10 mg) bupivacaine + 0.1 ml (100 mcg) morphine + 0.5 ml saline.
  Interventions: Procedure: Group morphine
- Group morfin+dexamethasone (Experimental): Group morfin+dexamethasone: Spinal anesthesia will be applied to patients who will undergo a caesarean section using a combination of 2 ml (10 mg) bupivacaine + 0.1 ml (100 mcg) morphine + 0.5 ml (2 mg) dexamethasone.
  Interventions: Procedure: Group morfin+dexamethasone

INTERVENTIONS:
Procedure: Group morphine — Group Morphine: Spinal anesthesia will be applied to patients who will undergo caesarean section using a combination of 2 ml (10 mg) bupivacaine + 0.1 ml (100 mcg) morphine + 0.5 ml saline
  Other Names: Group I
  Arms: Group morfin
Procedure: Group morfin+dexamethasone — Group morfin+dexamethasone: Spinal anesthesia will be applied to patients who will undergo a caesarean section using a combination of 2 ml (10 mg) bupivacaine + 0.1 ml (100 mcg) morphine + 0.5 ml (2 mg) dexamethasone
  Other Names: Group II
  Arms: Group morfin+dexamethasone

SUMMARY:
The Efficacy of Intrathecal Morphine Versus Intrathecal Morphine+Dexamethasone Combination added to bupivacaine in elective cesarean section under spinal anesthesia

DETAILED DESCRIPTION:
The study will be designed as a double-blind, randomized clinical trial and will be conducted following approval by the local ethics committee. A total of 120 patients, aged 18-40 years, with an ASA physical status of II and scheduled for elective cesarean section, will be included. All patients will undergo standard preparation for spinal anesthesia. Two large-bore intravenous lines will be inserted in each patient upon arrival in the operating room. Participants will be randomly assigned to one of two groups (n = 60 per group) using sealed opaque envelopes.

Group I (morphine group) will receive spinal anesthesia consisting of 2 mL (10 mg) bupivacaine, 0.1 mL (100 mcg) morphine, and 0.5 mL saline.

Group II (morphine+dexamethasone group) will receive a mixture of 2 mL (10 mg) bupivacaine, 0.1 mL (100 mcg) morphine, and 0.5 mL (2 mg) dexamethasone.

Intraoperative hemodynamic parameters (including age, height, and weight), ASA scores, postoperative complications (such as nausea, vomiting, and pruritus), and postoperative pain levels will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for caesarean sections
* Between 18-40 years
* ASA II group
* Those who will undergo spinal anesthesia
* Those between 35-40 weeks of pregnancy
* 1st and 2nd caesarean sections

Exclusion Criteria:

* Those who prefer general anesthesia
* Those who are outside the age range of 18-40
* Those who are ASA III and above
* Those with HT, DM, cardiac and respiratory diseases
* Preeclampsia, eclampsia, HELLP
* Those with a history of drug use that affects the cardiovascular system
* Placenta Previa, Placenta Acreta, Placenta Acreta Those with a history of antiemetic or antidepressant drug use

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea-vomiting | For 24 hours after surgery
  The incidence of postoperative nausea and vomiting will be scored from 0 to 3. No nausea or vomiting attacks will be graded as 0, a nausea attack that resolves without treatment will be graded as 1, recurrent nausea attacks that resolve with treatment will be graded as 2, and persistent nausea or vomiting attacks will be graded as 3.
Postoperative itching | For 24 hours after surgery
  The degree of pruritus will be assessed on a scale of 0 to 3, with 0 being categorized as no pruritus; 1 as mild pruritus; 2 as moderate pruritus; and 3 as severe pruritus.

SECONDARY OUTCOMES:
Intraoperative Mean Blood Pressure | Intraoperatively every 5 minutes
  Mean blood pressure will be measured every 5 minutes intraoperatively using a noninvasive method.
Intraoperative Heart Rate | Intraoperatively every 5 minutes
  Heart rate will be measured every 5 minutes intraoperatively using a noninvasive method

CONTACTS AND LOCATIONS:
Overall Officials: Nurettin KURT, Assoc.Prof, Principal Investigator — YüzüncüYıl

IPD SHARING:
Plan to Share IPD: Yes
Study protocol anda statistical analysis plan will be share with other researchers
Supporting Information: Study Protocol, SAP
Time Frame: 10 months
Access Criteria: The access can be provided via the e-mail addresses below dr.nurettinkurt@gmail.com

REFERENCES:
- [Background] Ankouni T, Kanawati S, El Khatib R, El Hassan J, Itani SE, Rajab O, Naja Z. Ondansetron versus ondansetron with dexamethasone to prevent intrathecal-morphine pruritus for caesarean patients: randomised double-blind trial. J Obstet Gynaecol. 2021 Oct;41(7):1080-1086. doi: 10.1080/01443615.2020.1852538. Epub 2021 Mar 2. PMID 33650930
- [Background] Nasiri A, Abutorabi SM, Sane S. Intrathecal dexamethasone-bupivacaine combination with bupivacaine alone in spinal anesthesia for cesarean delivery. Caspian J Intern Med. 2024 Summer;15(3):414-420. doi: 10.22088/cjim.15.3.414. PMID 39011433
- [Background] Ahmed SA, Lotfy HA, Mostafa TAH. The effect of adding dexmedetomidine or dexamethasone to bupivacaine-fentanyl mixture in spinal anesthesia for cesarean section. J Anaesthesiol Clin Pharmacol. 2024 Jan-Mar;40(1):82-89. doi: 10.4103/joacp.joacp_396_22. Epub 2024 Mar 14. PMID 38666154